CLINICAL TRIAL: NCT02860468
Title: To Determine the Metabolomics and Microbiome Changes After Cranberry Juice Consumption Among Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201601249
Record Dates: First submitted 2016-07-25; First posted 2016-08-09 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry juice consumption (Experimental): participants in this arm will be provided cranberry juice to consume for 21 days in total
  Interventions: Other: Cranberry juice
- Placebo juice consumption (Placebo Comparator): participants in this arm will be provided placebo juice to consume for 21 days in total
  Interventions: Other: Placebo juice

INTERVENTIONS:
Other: Cranberry juice — cranberry juice cocktail provided by Ocean Spray Cranberries, Inc.
  Arms: Cranberry juice consumption
Other: Placebo juice — apple juice added with flavor and colorants provided by Ocean Spray Cranberries, Inc.
  Arms: Placebo juice consumption

SUMMARY:
The compliance of participants in cranberry related clinical trial is poor due to the bitterness and astringency of cranberry products. There is a pressing need for an effective approach to verify participant compliance. The PLS-DA (Partial Least Squares Discriminant Analysis) /OPLS-DA (Orthogonal Partial Least Squares Discriminant Analysis) models established from the investigator's previous study provide an opportunity to identify cranberry juice consumers. In this blinded, placebo-controlled, cross-over study, investigators hypothesize that the established statistical models of PLS-DA (Partial least squares discriminant analysis) /OPLS-DA (Orthogonal partial least squares discriminant analysis) can identify cranberry juice consumers and non-consumers by analyzing the metabolomic changes in blood and urine among young women. In order to further explore the function of cranberry, microbiome profile will also be compared between cranberry juice consumption and placebo consumption after long-term treatment. Another comparison of metabolomic changes between short-term treatment and long-term treatment will be made to further identify candidate biomarkers of cranberry consumption and explore the correlation between acute effects and chronic effects of cranberry.

DETAILED DESCRIPTION:
Consumption of cranberry juice has been related to the prevention of urinary tract infection. However, due to the bitterness and astringency of cranberry products, the compliance of participants in cranberry related clinical trial is poor, which makes it difficult to further study the function of cranberry juice. Accordingly, there is a pressing need for an effective approach to verify participant compliance. In the previous study, plasma and urinary metabolome in young women following cranberry juice consumption have been investigated using a global UHPLC (Ultra high-performance liquid chromatography) -Q-Orbitrap-HRMS (High-resolution mass spectrometry) approach. PLS-DA (Partial least squares discriminant analysis) analyses showed that both plasma and urinary metabolome in young women were altered following cranberry consumption compared to baseline and apple juice consumption. Cranberry juice consumption caused a greater excretion of both exogenous and endogenous metabolites. These metabolites have been identified as candidate biomarkers for cranberry juice consumption. The established PLS-DA (Partial least squares discriminant analysis) /OPLS-DA (Orthogonal partial least squares discriminant analysis) models provide an opportunity to identify cranberry juice consumers.

It is unknown whether cranberry juice consumption influences gut microbiota profile in human. But several studies suggested that a polyphenol-rich diet improves gut microbiota profile. The previous in vitro study with human gut microbiota indicated that microbial catabolism of A-type cranberry procyanidins produced metabolites with different profiles and structures compared with those from B-type procyanidins.

Understanding microbiome change in human gut will enable the investigators to correlate and explain metabolome changes in the urine and blood, and also will explain the health benefits of cranberries.

With all the samples will be collected in this study, the metabolomics changes between short-term cranberry juice treatment (3days) and long-term treatment (21days) can be compared. Since the urinary tract protection effects of cranberry juices are often associated with chronic consumption, more metabolomic changes are expected to be identified by a long-term study.

Research Plan:

Specific aim 1: Twenty (20) healthy female college students aged 18-29 with normal BMI (Body mass index) (18.5-25) and at least 110 pounds in weight will be recruited on UF (University of Florida) campus.

Advertisement will be in the form of flyers. Contact information of investigators will be included in the flyer. Questionnaire will be used to obtain information about subjects for prescreen. All participants will be received written and oral information regarding the natural and potential risks of the study.

Participants will be advised to avoid proanthocyanidins-rich foods including cranberries, blueberries, strawberries plum, raspberries, apple, grapes, grape seed extract, pycnogenol, red wine, tea, chocolate and other cocoa products or other cranberry based supplements from the beginning of 10-day (1st-9th ) run in period to the end of the study. Participants will be suggested to consume orange, watermelon, honey dew, cantaloupe for replacement. Urine and stool sample collection kits will be distributed to all participants and participants will be trained to use the collection kits. One fecal sample will be collected by participants during any day from the 7th to 9th day. On the 10th day morning, overnight fast urine sample will be self-collected and subjects will have blood sample drawn (2 tubes, 30mL total). Breakfast will be provided for participants after fasting blood sample collection. A trained and certified phlebotomist will be hired to draw blood. After blood drawn, each participant will consume 1 bottle (250mL) of cranberry or placebo juice and another 5 bottles of cranberry or placebo juice will be given to each subject to consume in the evening of the 10th day and in the morning and evening of the 11th and12th day. One fecal sample will also be collected during the 12th- 4th day. All subjects will return to the clinical unit in the morning of the 13th day with a self-collected overnight fast urine sample and blood samples will be collected 30-60min after participants consume 1 bottle of cranberry or placebo juice. Cranberry or placebo juice will be distributed to each of the subjects to consume in the evening of the 13th day and in the morning and evening during the 14th- 29th day. Appointment will be scheduled weekly or upon the request of participants during the 14th to 29th day. One fecal sample will be collected during the 29th to 31st day. In the morning of the 30th day, overnight fast urine sample will be self-collected and subjects will have blood sample drawn after consume cranberry juice or placebo. After 14-days washout period, participants will switch to the alternative regimen and repeat the protocol. All samples collected will be aliquoted and kept in -80°C. It's unlikely to happen, but if any subject has any serious adverse effect after juice consumption, participant will be removed from the study depending on her situation for safety concern.

Preparation of urine and plasma sample collected at the13th, 48th day (3 days later after cranberry juice/placebo consumption) will follow established protocols. LC-HRMS (Liquid chromatography - High-resolution mass spectrometry) data will be normalized and imported to SIMCA (Version 13.0.3, Umetrics, Umea, Sweden) to use previously established PLS-DA (Partial least squares discriminant analysis) /OPLS-DA (Orthogonal partial least squares discriminant analysis) models to blindly identify cranberry juice consumers. Results will be sent to Ocean Spray for verification.

Specific aim 2:

The baseline fecal samples and fecal sample collected around the 30th, 65th day (21 days later after cranberry juice/placebo consumption) will be analyzed for microbiome composition. Genomic microbial DNA will be extracted from stool samples using MoBlo Power soil DNA isolation kits.. Microbiota change in the gut will be correlated with metabolome changes in the urine using redundancy and discriminant analysis. Fecal mucin and IgA (Immunoglobulin A, indicators of intestinal barrier), short chain fatty acids and ammonia in the stool samples will be analyzed using specific assay kits or HPLC (High-performance liquid chromatography) method.

Specific aim 3:

Preparation of urine and plasma sample collected at the 30th, 65th day (21 days later after cranberry juice/placebo consumption) will follow established protocols. UHPLC (Ultra high-performance liquid chromatography) -Q-Orbitrap-HRMS (High-resolution mass spectrometry) analyses, Multivariate data processing and statistical analysis will be the same as the experiment process discussed in Specific aim 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal BMI (18.5-25)
* Body weight ≥110 pounds

Exclusion Criteria:

* Gastrointestinal disorders
* Urological diseases
* Metabolic disorders
* Smokers
* Pregnancy
* Previous use of antibiotics or probiotics.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-03-25 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
The correct rate of identifying cranberry consumers and non-cranberry consumers by previously established multivariate statistical models of PLS-DA/OPLS-DA combined with UHPLC-Q-Orbitrap-HRMS. | up to 6 months

SECONDARY OUTCOMES:
Number of healthier microbial community in the stool sample after short-term (3 days) and long-term (21 days) cranberry juice consumption. | 3 days and 21 days
The change in quantity of endogenous and exogenous metabolites in blood/urine after 3-day consumption and 21-day consumption of cranberry juice comparing to baseline blood/urine sample | 3 days and 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Gu, PhD, Principal Investigator — University of Florida
Locations (1):
- Food Science and human nutrition department at University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jepson R, Craig J, Williams G. Cranberry products and prevention of urinary tract infections. JAMA. 2013 Oct 2;310(13):1395-6. doi: 10.1001/jama.2013.277509. PMID 24084925
- [Background] Liu H, Garrett TJ, Tayyari F, Gu L. Profiling the metabolome changes caused by cranberry procyanidins in plasma of female rats using (1) H NMR and UHPLC-Q-Orbitrap-HRMS global metabolomics approaches. Mol Nutr Food Res. 2015 Nov;59(11):2107-18. doi: 10.1002/mnfr.201500236. Epub 2015 Sep 15. PMID 26264887
- [Background] Ou K, Sarnoski P, Schneider KR, Song K, Khoo C, Gu L. Microbial catabolism of procyanidins by human gut microbiota. Mol Nutr Food Res. 2014 Nov;58(11):2196-205. doi: 10.1002/mnfr.201400243. Epub 2014 Aug 22. PMID 25045165